CLINICAL TRIAL: NCT02723487
Title: Postoperative Analgesic Efficacy of Transversus Abdominis Plane Block by Bupivacaine With Two Different Concentrations in Pediatric Patient Undergoing Laparoscopic Surgery
Brief Title: Ultrasound Guided Transversus Abdominis Plane Block in Pediatric Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abdelrady S Ibrahim, MD (Other)
Responsible Party: Sponsor-Investigator, Abdelrady S Ibrahim, MD, Assistant professor of Anesthesia and Intensive care, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17100390
Record Dates: First submitted 2016-03-14; First posted 2016-03-30 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Postoperative Pain
Keywords: TAP block; pediatric; Laparoscopic; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (No Intervention): Control
- Group B (Active Comparator): patients will receive bilateral ultrasound guided TAP block using bupivacaine (0.125%), 0.5 ml/kg on each side.
  Interventions: Drug: Bupivacaine 0.125%
- Group C (Active Comparator): patients will receive bilateral ultrasound guided TAP block using bupivacaine (0.25%), 0.5 ml/kg on each side.
  Interventions: Drug: Bupivacaine 0.25%

INTERVENTIONS:
Drug: Bupivacaine 0.125% — Patients will receive bilateral Transversus Abdominis Plane Block guided by ultrasound device using bupivacaine (Marcaine, 0.125%), 0.5 ml/kg on each side.
  Other Names: Plain marcaine
  Arms: Group B
Drug: Bupivacaine 0.25% — Patients will receive bilateral Transversus Abdominis Plane Block guided by ultrasound device using bupivacaine (Marcaine, 0.25%), 0.5 ml/kg on each side.
  Other Names: Plain marcaine
  Arms: Group C

SUMMARY:
The primary objective of this study is to assess differences in postoperative pain experienced by pediatric patients having transversus abdominis plane block block with bupivacaine (0.125% and 0.25%) compared with control group will receive conventional iv analgesia after Laparoscopic surgery.

DETAILED DESCRIPTION:
A prospective randomized controlled double blind study using a computer generated randomization will be conducted in Assiut University Hospitals and carried on 60 pediatric patients undergoing laparoscopic surgery under general anesthesia.

After induction of general anesthesia and endotracheal intubation, patients in group B and group C will be placed in the supine position and transversus abdominis plane block will be performed under ultrasound guidance. After skin preparation, the linear ultrasound probe connected to a portable ultrasound unit will be placed in the axial plane across the mid-axillary line midway between the costal margin and the highest point of iliac crest. needle attached to a syringe filled with the Local anesthetic solution will be inserted until it reaches the plane between the internal oblique and transversus abdominis muscles.

After careful aspiration to exclude vascular puncture, injection of bupivacaine will be performed leading to separation between the internal oblique and the transversus abdominis muscles which will appear as a hypoechoic space on ultrasound. This procedure will be repeated on the opposite side .

Laparoscopic procedure will be started 20 minutes after completion of bilateral transversus abdominis plane block and 0.01 mg/kg iv atropine will be given before pneumoperitonem. Intra abdominal pressure will be maintained at 10-12 mmHg.

The use of opioids during the procedure will based on the cardiovascular response to stimulation; a heart rate increase of 20% from baseline will be interpreted as insufficient analgesia and will be treated with fentanyl in doses of 1mcg / kg.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II physical status patients.
* Genders Eligible for Study :male.
* All children scheduled for laparoscopic surgery between the ages of 1and 5 years.
* Duration of Laparoscopic procedure not exceeding 90 minutes.
* Written informed consent from parent of guardian .

Exclusion Criteria:

* Sensitivities to local anesthetics.
* Significant renal, liver, or cardiac disease.
* Surgery requiring an open procedure

Ages: 1 Year to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — According to type of surgery laparoscopic undescended testis
Enrollment: 60 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
pain score | 12 hours postoperative
  Children's Hospital Eastern Ontario Pain Scale

SECONDARY OUTCOMES:
Total intraoperative fentanyl consumption | 12 hours postoperative
  Microgram (ug)
number of participants with incidence of nausea | 12 hours postoperative
  number of patients
number of participants with incidence of hematoma | 12 hours postoperative
  number of patients
number of participants with incidence of infection | 12 hours postoperative
  number of patients
Total postoperative paracetamol consumption | 12 hours postoperative
  Milligram (mg)
Number of participants with incidence of vomiting | 12 hours postoperative
  number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrady s Ibrahim, MD, Principal Investigator — Assistant profossor
Locations (1):
- Assiut university faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Long JB, Birmingham PK, De Oliveira GS Jr, Schaldenbrand KM, Suresh S. Transversus abdominis plane block in children: a multicenter safety analysis of 1994 cases from the PRAN (Pediatric Regional Anesthesia Network) database. Anesth Analg. 2014 Aug;119(2):395-399. doi: 10.1213/ANE.0000000000000284. PMID 24918899